CLINICAL TRIAL: NCT02546102
Title: A Phase 3 Randomized Double-blind, Controlled Study of ICT-107 With Maintenance Temozolomide (TMZ) in Newly Diagnosed Glioblastoma Following Resection and Concomitant TMZ Chemoradiotherapy
Brief Title: Phase 3 Randomized, Double-blind, Controlled Study of ICT-107 in Glioblastoma
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Company is discussing with FDA to reinitiate the trial now.
Sponsor: Precision Life Sciences Group (Industry)
Collaborators: Medelis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICT-107-301
Record Dates: First submitted 2015-09-07; First posted 2015-09-10 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Arm 1 will receive ICT-107 in combination with the standard of care, temozolomide (TMZ). ICT-107 will be given once a week for 4 weeks in the induction phase. During the maintenance phase, ICT-107 will be given monthly for the 11 months after induction and once every 6 months thereafter until depletion of supply or confirmation of progressive disease (PD). Administration is intradermal in axilla.
  Interventions: Biological: ICT-107
- 2 (Placebo Comparator): Arm 2 will receive TMZ with a blinded control. Control will be given once a week for 4 weeks in the induction phase. During the maintenance phase, Control will be given monthly for the 11 months after induction and once every 6 months thereafter until depletion of supply or confirmation of progressive disease (PD). Administration is intradermal in axilla.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ICT-107 — Autologous dendritic cells pulsed with peptides associated with tumor antigens
  Arms: 1
Biological: Placebo — Control, autologous monocytes-enriched PBMC.
  Arms: 2

SUMMARY:
ICT-107 consists of dendritic cells, prepared from autologous mononuclear cells that are pulsed with six synthetic peptides that were derived from tumor associated antigens (TAA) present on glioblastoma tumor cells. This is a Phase 3 study to evaluate ICT-107 in patients with newly diagnosed glioblastoma. Subjects will be randomized to receive standard of care chemoradiation (temozolomide (TMZ) with either ICT-107 or a blinded control. Reinfusion with the pulsed dendritic cells should stimulate cytotoxic T cells to specifically target glioblastoma tumour cells.

DETAILED DESCRIPTION:
This is a double blind Phase III study where eligible subjects are randomized into two treatment arms following the SOC primary treatment with chemoradiation: Arm 1 will receive ICT-107 in combination with the standard of care, temozolomide (TMZ), Arm 2 will receive TMZ with a blinded control. A 1:1 randomization will be employed, where ARM 1 will receive ICT-107 and Arm 2 will receive placebo control. All subjects must be HLA-A2+. All subjects must have glioblastoma tissue that has tumor assessment for MGMT methylation status prior to randomization (for stratification). Subjects will have had tumor resection and magnetic resonance imaging (MRI) prior to enrollment into the study. After signing of written informed consent and any required privacy compliance forms and screening, enrolled subjects will undergo large volume apheresis at the study site for collection of PBMCs. Apheresis product will be sent to the manufacturing site where both active therapy (ICT-107) and control will be prepared for each subject prior to randomization The study period consists of 4 time periods; a 6-week Post-Surgery Standard of Care Treatment Phase where subjects receive radiotherapy and TMZ; TMZ and radiation to be initiated no more than 8 weeks after surgical resection of glioblastoma; a Rest Period of no more than 14 days where subjects are reassessed for eligibility, and then randomized; a 4 week Induction Phase where study therapy (ICT-107 or Control) is given weekly; followed by a Maintenance Phase where study therapy is given monthly for 11 months, and then every 6 months until either progression, withdrawal from the study, death, or the supply of autologous study therapy is exhausted. Randomized subjects will receive 4 weekly administrations of subject-specific study therapy (ICT-107 or Control) during the Induction Phase. No TMZ will be given during the 4 week Induction Phase. Each study therapy injection will be delivered intradermally (axilla).

The Maintenance Phase will consist of administration of subject-specific study therapy monthly for 11 months after the Induction Phase (for a total of 15 injections over 12 months during the Induction and Maintenance Phases), and then every 6 mos. thereafter until depletion or confirmation of progressive disease (PD). During the Maintenance Phase (where ICT-107 or control are given monthly), the administration of TMZ and subject specific study therapy or control will be separated in time by approximately 2 weeks (see Section 9.1.4). Pre-treatment, treatment and assessment schedules will be the same for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and sign the study specific informed consent
2. Subjects must be in primary remission
3. Subjects should have < 1 cm3 disease by MRI within the previous 4 weeks (by central read)
4. Subjects must be HLA-A2 positive by central lab
5. Subjects must have adequate renal, hepatic and bone marrow function based on screening laboratory assessments. Baseline hematologic studies and chemistry and coagulation profiles must meet the following criteria:

   1. Hemoglobin (Hgb) > 8 g/dL
   2. Absolute Neutrophil Count (ANC) > 1000/mm3
   3. Platelet count > 100,000/mm3
   4. Blood Urea Nitrogen (BUN) < 30 mg/dL
   5. Creatinine < 2 mg/dL
   6. Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2 x upper limit of normal (ULN)
   7. Prothrombin Time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6x unless therapeutically warranted
6. Subjects must use effective contraceptive methods during the study and for three months following the last dose of study product, if of reproductive age and still retain fertility potential.
7. Subjects must have at least one positive DTH skin response (more than 5 mm) to test item challenge prior to randomization.

Exclusion Criteria:

1. Subjects receiving investigational study drug for any indication or immunological-based treatment for any reason (Filgrastim may be used for prevention of severe neutropenia).
2. Subjects with glioblastoma mutated IDH by Immunohistochemistry (IHC)
3. Subjects with concurrent conditions that would jeopardize the safety of the subject or compliance with the protocol.
4. Subjects with a history of chronic or acute hepatitis C or B infection.
5. Subjects require or are likely to require more than a 2-week course of corticosteroids for intercurrent illness. Subjects must have completed the course of corticosteroids at the time of apheresis to meet eligibility.
6. Subjects have any acute infection that requires specific therapy. Acute therapy must have been completed within seven days prior to study enrollment.
7. Subjects with active other malignancy diagnosed in the past 3 years (excepting in situ tumors)
8. Subjects known to be pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 46 months
  Overall survival (OS) of subjects treated with ICT-107 and standard of care (radiation (RT) and TMZ) vs. placebo control and standard of care (RT and TMZ)

SECONDARY OUTCOMES:
Overall survival in patients with unmethylated MGMT tumors | 46 months
  OS of subjects with unmethylated MGMT (O6-methylguanine-DNA methyltransferase) tumors treated with ICT-107 and standard of care vs. control and standard of care
Overall survival in patients with methylated MGMT (O6-methylguanine-DNA methyltransferase) tumors | 46 months
  OS of subjects with methylated MGMT tumors treated with ICT-107 and standard of care vs. control and standard of care.
Progression-free survival | 46 months
  Progression-free survival (PFS) of subjects treated with ICT-107 and standard of care vs. control and standard of care
Type and frequency of treatment emergent adverse events | 46 months
  Compare the type and frequency of treatment emergent adverse events of ICT-107 vs. control treatment groups

CONTACTS AND LOCATIONS:
Locations (65):
- United States (58):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dignity Health - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - City of Hope Cancer Center, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Irvine Chao Family Cancer Center, Orange, California
  - Kaiser Permanente, Redwood City, California
  - Kaiser Permanente, Sacramento, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Delray Medical Center, Boca Raton, Florida
  - Boca Raton Regional Hospital Lynn Cancer Institute, Boca Raton, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - John Nasseff Neuroscience Institute, Minneapolis, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - JFK New Jersey Neuroscience Institute, Edison, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - North Shore University Hospital, Lake Success, New York
  - Perlmutter Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weil Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State College of Medicine Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Pavilion, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Cancer Institute, Knoxville, Tennessee
  - Texas Oncology, Austin, Texas
  - Baylor Health Charles Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center Memorial Hermann Hospital, Houston, Texas
  - CTRC at UTHSCSA, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Ivy Center for Advanced Brain Tumor Treatment Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Austria (3):
  - Medical University Innsbruck, Dept. of Neurology, Innsbruck
  - Kepler Universitätsklinikum, Neuromed Campus, Linz
  - University Clinic for Neurology, Salzburg
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
  - CHUS Service de Neurochirurgie, Sherbrooke, Quebec

REFERENCES:
- [Result] Phuphanich S, Wheeler CJ, Rudnick JD, Mazer M, Wang H, Nuno MA, Richardson JE, Fan X, Ji J, Chu RM, Bender JG, Hawkins ES, Patil CG, Black KL, Yu JS. Phase I trial of a multi-epitope-pulsed dendritic cell vaccine for patients with newly diagnosed glioblastoma. Cancer Immunol Immunother. 2013 Jan;62(1):125-35. doi: 10.1007/s00262-012-1319-0. Epub 2012 Jul 31. PMID 22847020